CLINICAL TRIAL: NCT01339390
Title: MOVE OUT: A Partnership With Veterans Groups to Enhance Weight Management in VHA
Brief Title: MOVE OUT: A Partnership With Veterans Groups to Enhance Weight Management in the Veterans Health Administration (VHA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The American Legion Department of Wisconsin (Other); Veterans Of Foreign Wars Of The United States Department Of Wisconsin (Other); All Saints Catholic Church, Milwaukee (Unknown); Three Holy Women Catholic Parish (Unknown); Veterans 76 Ltd. (Other); Dryhootch of America, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 10-327; 1I01HX000562-01A1 (NIH)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Overweight; Hypertension; Diabetes Mellitus
Keywords: Obesity; Veteran; Self Care; Patient Education; Peer Group
MeSH Terms: conditions — Obesity; Overweight; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: MOVE OUT (Experimental): The MOVE OUT intervention builds on the high quality information provided by the nationally-developed MOVE! program by adding 1) peer support; 2) convenient local access to educational sessions, which allows the material to be delivered in smaller, more easily retained aliquots; 3) convenient local exercise opportunities; and 4) open-ended availability of both education and exercise support.
  Interventions: Behavioral: MOVE OUT
- Arm 2: MOVE! (Active Comparator): As part of routine care at the ZVAMC, all patients who are eligible for the present study are identified by a "clinical reminder." This reminder prompts the primary care provider (PCP) to determine if the person would benefit from a weight loss program, and to refer them to MOVE! if they and the patient agree that it would be beneficial. The MOVE! program in Milwaukee can be tailored by the patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
  Interventions: Behavioral: MOVE!

INTERVENTIONS:
Behavioral: MOVE OUT — The MOVE OUT intervention builds on the high quality information provided by the nationally-developed MOVE program by adding 1) peer support; 2) convenient local access to educational sessions, which allows the material to be delivered in smaller, more easily retained aliquots; 3) convenient local exercise opportunities; and 4) open-ended availability of both education and exercise support.
  Arms: Arm 1: MOVE OUT
Behavioral: MOVE! — As part of routine care at the ZVAMC, all patients who are eligible for the present study are identified by a "clinical reminder." This reminder prompts the PCP to determine if the person would benefit from a weight loss program, and to refer them to MOVE if they and the patient agree that it would be beneficial. The MOVE program in Milwaukee can be tailored by the patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
  Arms: Arm 2: MOVE!

SUMMARY:
Obesity has been linked to several serious medical conditions, including high blood pressure, diabetes, and poor cholesterol levels. For this reason, obesity is likely the most important single contributor to cardiovascular mortality in the United States. Fortunately, intensive weight management programs are an effective treatment for obesity. Such programs help people lose weight and improve their measures of cardiac risk. In response to the growing numbers of obese Veterans being treated at Veterans Health Administration (VHA) facilities, the VHA developed the MOVE! Program. Veterans who commit to MOVE! and participate actively do lose weight. Unfortunately, MOVE!, like other weight management programs, requires its participants to attend classes and to exercise, often at locations and times that are inconvenient. The investigators propose to make it easier for eligible patients at the Zablocki Veterans Affairs Medical Center (ZVAMC) to participate by offering MOVE-style classes and exercise groups at a variety of locations, days, and times. The investigators' program-MOVE OUT-may provide a model for VHA to use nationwide.

DETAILED DESCRIPTION:
Background: Obesity increases the prevalence and severity of cardiovascular risk factors such as hypertension, diabetes, and metabolic syndrome. It is also a leading contributor to cancer and osteoarthritis. Obesity and overweight are highly prevalent among VHA patients: As with the general population, over two-thirds of VHA users are either overweight or obese. There is good evidence that intensive weight reduction programs can have a modest-but clinically significant-impact on weight. VHA has developed a comprehensive weight management program known as MOVE! to address obesity among its patients. MOVE! evaluations to date have demonstrated success in helping Veterans lose weight, but participation is low. In the investigators' preliminary work, the investigators found that the timing (daytime) and location (ZVAMC) of MOVE! activities were viewed by eligible patients as barriers to participation. In addition, previous research has often demonstrated significant rebound in weight at the end of formal program activities, which may be mitigated if there is a convenient place for ongoing weight monitoring and healthy activities with peers.

Objectives: The overall goal of the project is to increase participation in the ZVAMC MOVE! program by implementing an innovative community-based program known as MOVE OUT. MOVE OUT will incorporate the key elements of the proven MOVE! program (education, peer support, and planned physical activity), but in settings closer to the homes of eligible Zablocki patients. The investigators have the following objectives:

1. To reduce the mean weight of high-risk overweight or obese Veterans who receive primary care at ZVAMC.
2. To improve the physical activity and diet of high-risk overweight or obese Veterans who receive primary care at ZVAMC.
3. To demonstrate that an innovative community-based program can increase the proportion of ZVAMC users who participate actively in a moderately intensive weight management program as recommended by the National Institutes of Health Consensus Conference on Obesity.

Methods: The investigators will use a cluster randomized trial design. The investigators will allocate groups of eligible Veterans from ZVAMC to either a MOVE OUT invitation or a standard MOVE! invitation. The investigators will use clinically gathered weight data to determine overall rates of weight loss in the randomly assigned Veterans. In addition, the investigators will recruit a sample of Veterans from each randomized group to participate in a study of the effectiveness of the weight management program to which they are assigned. The investigators will use established methods to assess changes in diet, exercise and attitude, as well as physiologic outcomes including weight, blood pressure, Hemoglobin A1c, and lipid values. The investigators will use qualitative methods to learn what aspects of the two programs are most effective.

Impact: The investigators will demonstrate that VHA can deliver effective weight management services in a community-based fashion. If this study finds that such a delivery approach leads to an increased number of at-risk Veterans participating in weight control programs, it will guide program design throughout VHA. Although weight management is particularly well suited to a disseminated delivery model, lessons learned from this research are likely to help VHA improve its ability to help patients self-manage a variety of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Visit to ZVAMC primary provider within 3 months
* BMI >= 30 OR BMI >= 25 and Hypertension or Diabetes Mellitus
* No scheduled appointment for a MOVE program clinic
* Age <= 75 years
* Live in targeted geographic region

Exclusion Criteria:

* None

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3169 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Whittle, MD MPH, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: MOVE!: As part of routine care, all patients who are eligible for the present study are identified by a "clinical reminder." This prompts the primary care provider (PCP) to determine if the person would benefit from a weight loss program, and to refer them to MOVE! if they and the patient agree that it would be beneficial. The MOVE! program in Milwaukee can be tailored by patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
  MOVE!: As part of routine care, all patients who are eligible for the present study are identified by a "clinical reminder." This reminder prompts the PCP to determine if the person would benefit from a weight loss program, and to refer them to MOVE! if they and the patient agree that it would be beneficial. The MOVE! program in Milwaukee can be tailored by the patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
Period: Overall Study
Arm/Group | Arm 1: MOVE OUT | Arm 2: MOVE!
Started | 1571 | 1598
Completed | 1414 | 1442
Not Completed | 157 | 156
Not completed — Death | 32 | 29
Not completed — Lost to Follow-up | 125 | 127

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: MOVE OUT: The MOVE OUT intervention builds on the high quality information provided by the nationally-developed MOVE program by adding 1) peer support; 2) convenient local access to educational sessions, which allows the material to be delivered in smaller, more easily retained aliquots; 3) convenient local exercise opportunities; and 4) open-ended availability of both education and exercise support.
  MOVE OUT: The MOVE OUT intervention builds on the high quality information provided by the nationally-developed MOVE program by adding 1) peer support; 2) convenient local access to educational sessions, which allows the material to be delivered in smaller, more easily retained aliquots; 3) convenient local exercise opportunities; and 4) open-ended availability of both education and exercise support.
- Arm 2: MOVE!: As part of routine care at the ZVAMC, all patients who are eligible for the present study are identified by a "clinical reminder." This reminder prompts the PCP to determine if the person would benefit from a weight loss program, and to refer them to MOVE if they and the patient agree that it would be beneficial. The MOVE program in Milwaukee can be tailored by the patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
  MOVE!: As part of routine care at the ZVAMC, all patients who are eligible for the present study are identified by a "clinical reminder." This reminder prompts the PCP to determine if the person would benefit from a weight loss program, and to refer them to MOVE if they and the patient agree that it would be beneficial. The MOVE program in Milwaukee can be tailored by the patient and PCP, but includes dietitian assessment, education, weekly weigh-ins, follow-up classes, and exercise programs.
- Total: Total of all reporting groups
Arm/Group | Arm 1: MOVE OUT | Arm 2: MOVE! | Total
Number analyzed (Participants) | 1571 | 1598 | 3169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1021 | 1028 | 2049
  >=65 years | 550 | 570 | 1120
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.26 (10.8) | 59.80 (10.4) | 59.54 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 54 | 120
  Male | 1505 | 1544 | 3049
Region of Enrollment [Number; unit: participants]
  United States | 1571 | 1598 | 3169
Weight [Mean (Standard Deviation); unit: pounds] | 230.16 (43.82) | 229.01 (42.74) | 229.58 (43.28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight (From Baseline)
Description: Weight as recorded in the medical record during a 6-month period around the follow-up point.
Time Frame: Measured at 12 and 24 months
Population: For the analysis, we included those lost to follow up by using the last observation carried forward to impute missing values
Measure: Least Squares Mean (Standard Deviation); unit: Pounds
Arm/Group | Arm 1: MOVE OUT | Arm 2: MOVE!
Number analyzed (Participants) | 1571 | 1598
Pounds
  12 months | -0.71 (12.04) | -0.31 (12.49)
  24 months | -1.64 (15.34) | -1.06 (15.22)
Statistical Analysis 1: Comparison: Arm 1: MOVE OUT vs Arm 2: MOVE!; This is the analysis at 12 months, comparing the change in weight from 12 months to baseline in our Move Out (arm 1) vs Move (arm 2) groups; Test type: Superiority or Other; p = 0.4937, t-test, 2 sided — calculated after fitting the data to a repeated measures mixed model to control for repeated subject and random site and group effects; accounted for repeated measures and random effects; Mean Difference (Final Values) = 0.3941, 95% CI 2-sided [-.7347 to 1.5229], Standard Error of Mean 0.5759 — The difference is expressed as the Move (arm 2) group minus the Move Out (arm 1) group
Statistical Analysis 2: Comparison: Arm 1: MOVE OUT vs Arm 2: MOVE!; This is the analysis at 24 months, comparing the change in weight from 24 months to baseline in our Move Out (arm 1) vs Move (arm 2) groups; Test type: Superiority or Other; p = 0.3062, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; accounted for repeated measures and random effects; Mean Difference (Final Values) = 0.5893, 95% CI 2-sided [-0.5395 to 1.7181], Standard Error of Mean 0.5759 — The difference is expressed as the Move (arm 2) group minus the Move Out (arm 1) group

ADVERSE EVENTS:
Time Frame: For each cohort, we followed them passively for two years.
Description: This was done using only the electronic health record. We made no provision for identifying specific adverse events, but did record mortality. this was identified using the VA mortality data.
Arm/Group | Arm 1: MOVE OUT | Arm 2: MOVE!
Serious Adverse Events (participants affected / at risk) | 32/1571 | 29/1598
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MOVE OUT (N=1571) | Arm 2: MOVE! (N=1598)
Death at 12 months (General disorders) | 7 | 6 — Mortality as ascertained by VA reporting system. This is believed to be very accurate for veterans who are actively involved in care in VHA.
Death at 24 months (General disorders) | 25 | 23 — Mortality as ascertained by VA reporting system. This is believed to be very accurate for veterans who are actively involved in care in VHA.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MOVE OUT (N=0) | Arm 2: MOVE! (N=0)
All others (General disorders) | 0 | 0 — We did not collect other adverse events in follow up, nor did we use the VA electronic health record (CPRS) to ascertain adverse events other than death

LIMITATIONS AND CAVEATS:
Because passive enrollment was allowed by our Institutional Review Board, we were able to enroll all eligible patients identified by our automated record review. However, very few of the veterans randomized to the intervention used the program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No